CLINICAL TRIAL: NCT04679415
Title: A Multi Center, Randomized, Double-blind, Parallel Design, Phase 2 Study to Evaluate the Efficacy and Safety of hzVSFv13 Compared to Standard of Care After Intravenous (IV) Administration With Add-on Standard of Care in COVID-19 Moderate to Severe Patients
Brief Title: Efficacy and Safety of hzVSF-v13 in Moderate to Severe Patients With COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImmuneMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: hzVSF_v13-0007
Record Dates: First submitted 2020-12-21; First posted 2020-12-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care + hzVSF-v13 200 mg at D1, hzVSF-v13 100mg at D3 and D7 IV (Experimental): Drug: hzVSF-v13 Dosage form: hzVSF-v13 40mg/mL in a 5mL vial Frequency: Dose at Day 1, 3, 7 Other names: a humanized monoclonal antibody (mAb)
  Interventions: Drug: hzVSF-v13
- Standard of care + hzVSF-v13 400 mg at D1, hzVSF-v13 200mg at D3 and D7 IV (Experimental): Drug: hzVSF-v13 Dosage form: hzVSF-v13 40mg/mL in a 5mL vial Frequency: Dose at Day 1, 3, 7 Other names: a humanized monoclonal antibody (mAb)
  Interventions: Drug: hzVSF-v13
- Standard of care + 3 doses of the placebo (normal saline) IV (Placebo Comparator): Drug: Placebo (Normal saline solution) Dosage form: 0.9% NaCl Solution Frequency Frequency: Dose at Day 1, 3, 7 Other names: 0.9% Normal saline
  Interventions: Drug: Placebo (Normal saline solution)

INTERVENTIONS:
Drug: hzVSF-v13 — Dosage form: hzVSF-v13 40 mg/mL in a 5 mL vial Frequency: Dose at Day 1, 3, 7
  Other Names: a humanized monoclonal antibody (mAb)
  Arms: Standard of care + hzVSF-v13 200 mg at D1, hzVSF-v13 100mg at D3 and D7 IV; Standard of care + hzVSF-v13 400 mg at D1, hzVSF-v13 200mg at D3 and D7 IV
Drug: Placebo (Normal saline solution) — Dosage form: 0.9% NaCl Solution Frequency: Dose at Day 1, 3, 7
  Other Names: 0.9% Normal saline
  Arms: Standard of care + 3 doses of the placebo (normal saline) IV

SUMMARY:
Explore the efficacy and confirm the safety of the concomitant administration of the standard of care and hzVSF-v13 in patients with COVID-19 infection

DETAILED DESCRIPTION:
Multi center, Randomized, Double-blind, Parallel group, Phase 2 clinical study

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged at least 18 years at screening
2. Those who have been admitted or scheduled to be admitted due to a diagnosis with moderate to severe COVID-19 by RT-PCR test within 4 days prior to screening
3. Patients whose findings of COVID-19 pneumonia have been confirmed by radiographic tests (CT and X-ray) at screening (e.g., ground glass opacity (GGO), crazy-paving pattern, or consolidation)
4. Those who fall under the following at screening:

   * Patients identified as moderate Oxygen saturation in the atmosphere (SpO2) ≥ 93% (respiratory rate ≥20/min or pulse rate ≥90 beats/min secondarily)
   * Patients identified as severe Oxygen saturation in the atmosphere (SpO2) < 93% with (respiratory rate ≥30/min or pulse rate ≥125 beats/min secondarily)
5. Those who have voluntarily provided a written consent to participate in this clinical study

Exclusion Criteria:

1. Individuals with a clinically significant history of hypersensitivity reactions to the components of hzVSF-v13, drugs containing components of the same class, or other drugs (aspirin, non-steroidal anti-inflammatory drugs, antibiotics, etc.)
2. Patients with pneumonia other than due to the novel coronavirus (SARS-CoV-2) infection (e.g., influenza virus pneumonia, bacterial pneumonia, and fungal pneumonia)
3. Patients with severe heart failure (NYHA Class III or higher)
4. Pregnant women
5. Men and women of childbearing potential who are planning to become pregnant or do not agree to use one or more of the clinically appropriate methods of contraception below from the first day until 120 days after the last day of investigational product administration Surgical infertility (e.g., bilateral tubal ligation, vasectomy) Hormonal contraceptives (implantable form, patch, oral administration) Double-barrier method (concomitant use of two of the following: IUD, male or female condom used with spermicide, contraceptive diaphragm, contraceptive sponge, cervical cap)

   Periodic abstinence (e.g., calendar, ovulation date, basal body temperature, post-ovulation methods) and coitus interruptus are not permitted as appropriate contraceptive methods,and effective contraceptive methods must be kept being used during the course of the clinical study.
6. Those who are scheduled to have organ transplantation
7. Those who have laboratory test results that fall under the following values at screening ALT or AST ≥5 times the upper limit of normal (ULN) eGFR < 30 mL/min/1.73m2 platelets < 50,000/mm3
8. Those who have a positive result for serology (hepatitis B, human immunodeficiency virus [HIV], and hepatitis C tests) at screening
9. Those who received other investigational products within 30 days prior to the screening visit
10. Others who have been determined to be ineligible to participate in the clinical study according to the investigator's medical opinion, or subject who will/planned to be transferred to other hospital within study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Clinical failure rate at Day 28 | Day 28
  The clinical failure rate is defined at Day 28 if patient reported any of
  * Death
  * Respiratory failure (patient is intubated)
  * Patient is in the Intensive Care Unit (ICU)

SECONDARY OUTCOMES:
Changes from baseline in the clinical improvement score on an 8-point scale at Day 7, Day 14, and Day 28 | Day 7, Day 14, Day 28
  Descriptive statistics for the changes from baseline in the clinical improvement score on an 8-point scale at Day 7, Day 14, and Day 28 shall be presented for each treatment group, and a two-sample t-test or the Wilcoxon ranksum test shall be performed depending on whether the normality assumption is satisfied in order to test differences of each study group compared to the control group.
Time to discontinuation of oxygen therapy after investigational product administration | Day 28
  The Kaplan-Meier curves for the time to discontinuation of oxygen therapy after investigational product administration shall be presented, and the median time and 95% confidence interval will be presented by treatment group. In addition, a log-rank test shall be performed, if necessary, to test differences of each study group compared to the control group.
Time to recovery* after investigational product administration (days) | Day 28
  * 0 to 3 points in the clinical improvement score on an 8-point scale The Kaplan-Meier curves for the time to recovery after investigational product administration shall be presented, and the median time and 95% confidence interval will be presented by treatment group. In addition, a log-rank test shall be performed, if necessary, to test differences of each study group compared to the control group.
Time to Clinical Improvement from randomization to clinical improvement (2 points decreased from the baseline score) (days) | Day 28
  The Kaplan-Meier curves for the time to Clinical Improvement after randomization shall be presented, and the median time and 95% confidence interval will be presented by treatment group. In addition, a log-rank test shall be performed, if necessary, to test differences of each study group compared to the control group.
Changes from baseline in PaO2/FiO2 at Day 7, Day 14, Day 21, and Day 28 | Day 7, Day 14, Day 21, and Day 28
  Descriptive statistics for the changes from baseline in PaO2/FiO2 at Day 7, Day 14, Day 21, and Day 28 shall be presented for each treatment group, and a two-sample t-test or the Wilcoxon rank-sum test shall be performed depending on whether the normality assumption is satisfied in order to test differences of each study group compared to the control group.
Changes from baseline in the NEWS 2 score at Day 7, Day 14, Day 21, and Day 28 | Day 7, Day 14, Day 21, Day 28
  Descriptive statistics for the changes from baseline in the NEWS 2 score at Day 7, Day 14, Day 21, and Day 28 shall be presented for each treatment group, and a two-sample t-test or the Wilcoxon rank-sum test shall be performed depending on whether the normality assumption is satisfied in order to test differences of each study group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Prasenohadi Prasenohadi, phD, Principal Investigator — Rumah Sakit Umum Persahabatan
Locations (3):
- Indonesia (3):
  - Rumah Sakit Pusat Pertamina (include RSPP Extension Simprug), Jakarta, Jakarta Special Capital Region
  - Rumah Sakit Pasar Minggu, Jakarta, Jakarta Special Capital Region
  - Rumah Sakit Umum Persahabatan, Jakarta, Jakarta Special Capital Region

IPD SHARING:
Plan to Share IPD: No